CLINICAL TRIAL: NCT05368779
Title: Online Psychosocial Intervention for Nursing Students Who Experienced Intimate Partner Abuse in Turkey: A Randomized Controlled Trial
Brief Title: Online Psychosocial Intervention for Nursing Students Who Experienced Intimate Partner Abuse in Turkey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Hacer DEMIRKOL, Principal Investigator, Bozok University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 19-10T/43
Record Dates: First submitted 2022-04-27; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Violence, Sexual; Violence, Physical; Violence, Gender-Based; Violence; Post Traumatic Stress Disorder; Post Traumatic Growth, Psychological
MeSH Terms: conditions — Coitus; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based Psychosocial Intervention Group (Experimental): The internet-based psychosocial intervention, which was based on Social Learning Theory and Cognitive Behavioral Therapy techniques, was delivered individually and electronically to the participants in the experimental group in eight sessions, each lasting up to 120 minutes, using videoconferencing.
  Interventions: Behavioral: The internet-based psychosocial intervention
- Control Group (No Intervention): No intervention was applied to the participants in the control group.

INTERVENTIONS:
Behavioral: The internet-based psychosocial intervention — Participants were provided psychoeducation on intimate partner abuse, psychological trauma, Social Learning Theory, and Cognitive Behavioral Therapy methods. Intimate partner abuse and psychological trauma were discussed in the context of sociocultural factors. Cognitive Behavioral Therapy approaches were used to attempt to normalize intimate partner abuse, psychological trauma and their effects on participants. Participants were exposed to trauma gradually with record of sessions watching and imaginary exposure methods for reducing avoidance behaviours. Schemas, intermediate beliefs, and automatic thoughts of participants were studied using Cognitive Behavioral Therapy approaches and cognitive restructuring was fulfilled. The universality of mental pain, the meaning of life, the integrate trauma into life histories of participants, expectations for the future romantic relationships, and post traumatic growth were all discussed in accordance with the goals and values of participants.
  Arms: Internet-based Psychosocial Intervention Group

SUMMARY:
Intimate partner abuse is very common among university students. Post-traumatic stress disorder is one of the most serious mental diseases caused by intimate partner abuse.The purpose of this study was to assess the impact of an internet-based psychosocial intervention based on Social Learning Theory and Cognitive Behavioral Therapy approaches on post-traumatic stress and growth in student nurses who had experienced intimate partner abuse.

DETAILED DESCRIPTION:
Background: Intimate partner abuse is very common among university students. Post-traumatic stress disorder is one of the most serious mental diseases caused by intimate partner abuse. An intervention with evidence-based applications to post-traumatic stress caused by intimate partner abuse and posttraumatic growth, using web-based applications that young people are familiar with, is considered important in order to protect the physical-mental health of university students, to increase their academic success, and to ensure that they establish healthy intimate partner relationships in the future.

Objective: The purpose of this study was to assess the impact of an internet-based psychosocial intervention based on Social Learning Theory and Cognitive Behavioral Therapy approaches on post-traumatic stress and growth in student nurses who had experienced intimate partner abuse.

Methods: The randomized controlled study that did not use blinding employed a 2x5 split-plot design. The universe of the study consisted of 371 student nurses. Students who met the eligibility criteria were randomly assigned to one of the two groups: experimental (n=17) and control (n=18). The internet-based psychosocial intervention, which was based on Social Learning Theory and Cognitive Behavioral Therapy techniques, was delivered individually and electronically to the students in the experimental group in eight sessions, each lasting up to 120 minutes, using videoconferencing. The Impact of Events Scale-Revised (IES-R) and the Posttraumatic Growth Inventory (PGTI) were used to measure the outcomes at the pre-test, post-test, 1-month follow-up, 3-month follow-up, and 6-month follow-up.

Discussion: The internet-based psychosocial intervention was found to be effective in reducing post-traumatic stress and experiencing post-traumatic growth in student nurses who had been exposed to partner violence with these positive effects lasting for six months. This study is one of the first web-based randomized controlled studies to address post-traumatic stress and growth together in university students who were exposed to intimate partner violence. It is hoped that the results of the study will guide the research to be carried out in this context by internet intervention in the future.

* This research was carried out as part of the Ege University Institute of Health Sciences Psychiatric Nursing Doctoral Thesis.

Funding: No funding

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Must have access to a computer and internet
* Must able to read and understand the Turkish language
* Must experience intimate partner abuse
* Must break up with the abuse perpetrator intimate partner
* Must be on a current stable dose of psychiatric medication (for at least the last 3 months) or do not use psychiatric medication
* Must display symptoms of post-traumatic stress (must get a score of 24 or more in the Impact of Events Scale-Revised)

Exclusion Criteria:

* Have be currently married
* Have a high risk of suicide
* Have a psychotic symptom
* Have a dissociative symptom
* Have a risky alcohol and substance use
* Have a receive a non-drug psychiatric treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Pre-intervention post-traumatic stress levels of participants in the experimental and control groups | Pre-test (pre-internet-based psychosocial intervention)
  The post-traumatic stress levels of the participants in the experimental and control groups were measured by the Impact of Event Scale-Revised. Impact of Event Scale-Revised has a scoring range of 0 to 88. The cut-off point for post-traumatic stress disorder in the Turkish validity and reliability study of the scale was determined as 24 points. The level of post-traumatic stress increases as the score obtained from Impact of Event Scale-Revised increases.
Post-intervention post-traumatic stress levels of participants in the experimental and control groups | Post-test (immediately after the end of the internet-based psychosocial intervention)
  The post-traumatic stress levels of the participants in the experimental and control groups were measured by the Impact of Event Scale-Revised. Impact of Event Scale-Revised has a scoring range of 0 to 88. The cut-off point for post-traumatic stress disorder in the Turkish validity and reliability study of the scale was determined as 24 points. The level of post-traumatic stress increases as the score obtained from Impact of Event Scale-Revised increases.
1-month follow-up post-traumatic stress levels of participants in the experimental and control groups | 1-month follow-up (one month after internet-based psychosocial intervention)
  The post-traumatic stress levels of the participants in the experimental and control groups were measured by the Impact of Event Scale-Revised. Impact of Event Scale-Revised has a scoring range of 0 to 88. The cut-off point for post-traumatic stress disorder in the Turkish validity and reliability study of the scale was determined as 24 points. The level of post-traumatic stress increases as the score obtained from Impact of Event Scale-Revised increases.
3-month follow-up post-traumatic stress levels of participants in the experimental and control groups | 3-month follow-up (three month after internet-based psychosocial intervention)
  The post-traumatic stress levels of the participants in the experimental and control groups were measured by the Impact of Event Scale-Revised. Impact of Event Scale-Revised has a scoring range of 0 to 88. The cut-off point for post-traumatic stress disorder in the Turkish validity and reliability study of the scale was determined as 24 points. The level of post-traumatic stress increases as the score obtained from Impact of Event Scale-Revised increases.
6-month follow-up post-traumatic stress levels of participants in the experimental and control groups | 6-month follow-up (six month after internet-based psychosocial intervention)
  The post-traumatic stress levels of the participants in the experimental and control groups were measured by the Impact of Event Scale-Revised. Impact of Event Scale-Revised has a scoring range of 0 to 88. The cut-off point for post-traumatic stress disorder in the Turkish validity and reliability study of the scale was determined as 24 points. The level of post-traumatic stress increases as the score obtained from Impact of Event Scale-Revised increases.
Pre-intervention post-traumatic growth levels of participants in the experimental and control groups | Pre-test (pre-internet-based psychosocial intervention)
  The post-traumatic growth levels of the participants in the experimental and control groups were measured by the Posttraumatic Growth Inventory.Posttraumatic Growth Inventory has a scoring range of 0 to 105. The cut-off point for post-traumatic growth of the scale was accepted as 63 points. The level of post-traumatic growth increases as the score obtained from Posttraumatic Growth Inventory increases.
Post-intervention post-traumatic growth levels of participants in the experimental and control groups | Post-test (immediately after the end of the internet-based psychosocial intervention)
  The post-traumatic growth levels of the participants in the experimental and control groups were measured by the Posttraumatic Growth Inventory.Posttraumatic Growth Inventory has a scoring range of 0 to 105. The cut-off point for post-traumatic growth of the scale was accepted as 63 points. The level of post-traumatic growth increases as the score obtained from Posttraumatic Growth Inventory increases.
1-month follow-up post-traumatic growth levels of participants in the experimental and control groups | 1-month follow-up (one month after internet-based psychosocial intervention)
  The post-traumatic growth levels of the participants in the experimental and control groups were measured by the Posttraumatic Growth Inventory.Posttraumatic Growth Inventory has a scoring range of 0 to 105. The cut-off point for post-traumatic growth of the scale was accepted as 63 points. The level of post-traumatic growth increases as the score obtained from Posttraumatic Growth Inventory increases.
3-month follow-up post-traumatic growth levels of participants in the experimental and control groups | 3-month follow-up (three month after internet-based psychosocial intervention)
  The post-traumatic growth levels of the participants in the experimental and control groups were measured by the Posttraumatic Growth Inventory.Posttraumatic Growth Inventory has a scoring range of 0 to 105. The cut-off point for post-traumatic growth of the scale was accepted as 63 points. The level of post-traumatic growth increases as the score obtained from Posttraumatic Growth Inventory increases.
6-month follow-up post-traumatic growth levels of participants in the experimental and control groups | 6-month follow-up (six month after internet-based psychosocial intervention)
  The post-traumatic growth levels of the participants in the experimental and control groups were measured by the Posttraumatic Growth Inventory.Posttraumatic Growth Inventory has a scoring range of 0 to 105. The cut-off point for post-traumatic growth of the scale was accepted as 63 points. The level of post-traumatic growth increases as the score obtained from Posttraumatic Growth Inventory increases.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyda Dülgerler, Assoc. Prof., Principal Investigator — Ege University
Locations (1):
- Bozok University, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No